CLINICAL TRIAL: NCT04159519
Title: SHAMAL: A Multicentre, Randomised, Open-Label, Parallel-Group, Active-Controlled, Phase IV Study to Assess the Reduction of Daily Maintenance ICS/LABA Treatment Towards Anti-Inflammatory Reliever Treatment in Patients With Severe Eosinophilic Asthma Treated With Benralizumab
Brief Title: A Study to Assess the Reduction of Daily Maintenance ICS/LABA Treatment Towards Anti-Inflammatory Reliever Treatment in Patients With Severe Eosinophilic Asthma Treated With Benralizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3250C00072; 2019-001924-37 (EudraCT Number)
Record Dates: First submitted 2019-10-22; First posted 2019-11-12 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Asthma; Severe Eosinophilic Asthma
Keywords: Anti-Inflammatory; Reduction period; Inhaled corticosteroids; long-acting β2 agonist
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — Budesonide, Formoterol Fumarate Drug Combination; benralizumab; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment reduction arm (Experimental): Participants will receive Benralizumab 30 mg every 8 weeks (Q8W) during the study period, and high-dose Symbicort maintenance 400/12 μg ×2 inhalations BID + Ventolin (salbutamol 100 μg) reliever as needed (PRN), tapering to, medium-dose Symbicort 200/6 μg ×2 inhalations BID maintenance + Symbicort 200/6 μg reliever PRN, low dose Symbicort 200/6 μg x 1 inhalation BID maintenance + Symbicort 200/6 μg reliever PRN; or Symbicort 200/6 μg reliever only, as per tapering scheme and depending on the degree of asthma control). The reduction period in this arm lasted for 32 weeks.
  Interventions: Drug: Symbicort®; Drug: Fasenra®; Drug: Ventolin®
- Reference arm (Experimental): Participants will receive Benralizumab 30 mg Q8W + high-dose Symbicort® 400/12 μg maintenance ×2 inhalations BID + Ventolin® (salbutamol 100 μg) reliever PRN therapy. Eligible participants randomised to the reference arm continued on high-dose Symbicort® maintenance treatment and Ventolin® reliever treatment.
  Interventions: Drug: Symbicort®; Drug: Fasenra®; Drug: Ventolin®

INTERVENTIONS:
Drug: Symbicort® — Participants will receive Budesonide 400 μg/formoterol fumarate 12 μg per inhalation or Budesonide 200 μg/formoterol fumarate 6 μg per inhalation.
  Other Names: budesonide/formoterol
Drug: Fasenra® — Participants will receive Benralizumab 30 mg/mL, 1 mL fill volume via subcutaneous injection every 4 weeks for first 3 doses (prior to study inclusion), every 8 weeks thereafter.
  Other Names: benralizumab
Drug: Ventolin® — Participants will receive Salbutamol sulfate 100 μg per inhalation as needed.
  Other Names: salbutamol

SUMMARY:
This is a multicentre, randomised, open-label, parallel-group, active-controlled, phase IV study to assess the reduction of daily Symbicort® maintenance to anti-inflammatory reliever treatment only in participants with severe eosinophilic asthma on Fasenra® treatment, while maintaining asthma control.

DETAILED DESCRIPTION:
This study will be conducted at 24 study sites in 3-5 countries. The study duration for each participant will be approximately 52-56 weeks. Approximately 240 participants with severe eosinophilic asthma taking high-dose Inhaled corticosteroids/ long-acting β2-agonist (ICS/LABA) who have been treated for severe eosinophilic asthma with at least 3 consecutive doses of Fasenra® and have clinically responded since the start of Fasenra® treatment (defined for the purpose of this study as an Asthma control questionnaire-5 item (ACQ-5 score) <1.5 at Visit 1 and Visit 2b) will be enrolled into this open-label study. The study consists of a Screening Visit (Visit 1) and 4- to 8-week screening and run-in period (to align the randomisation study visit with the next Fasenra® injection), a reduction period of 32 weeks, and a 16-week maintenance period.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures.
2. Patient must be aged 18 years old or above at the time of consenting to study participation.
3. Documented current maintenance treatment with high-dose ICS/LABA.
4. ACQ-5 score <1.5 at Visit 1.
5. Treatment with Fasenra® for the indicated diagnosis of severe eosinophilic asthma and has received at least 3 consecutive doses (>8 weeks) prior to Visit 1.
6. Male or female.
7. Negative serum pregnancy test at Visit 1 for women of childbearing potential (WOCBP).
8. WOCBP must agree to use a highly effective method of birth control (confirmed by the Investigator) from randomisation throughout the study duration and within 12 weeks after the last dose of study treatment. Highly effective forms of birth control (those that can achieve a failure rate of less than 1% per year when used consistently and correctly) include:

   * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation-oral, intravaginal, or transdermal.
   * Progestogen-only hormonal contraception associated with inhibition of ovulation-oral, injectable, or implantable.
   * Intrauterine device (IUD).
   * Intrauterine hormone-releasing system (IUS).
   * Bilateral tubal occlusion.
   * Sexual abstinence, ie, refraining from heterosexual intercourse (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient).
   * Vasectomised sexual partner (provided that partner is the sole sexual partner of the WOCBP study patient and that the vasectomised partner has received medical assessment of the surgical success).

Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for ≥12 months prior to the planned date of randomisation without an alternative medical cause.

The following age-specific requirements apply:

* Women <50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and have follicle stimulating hormone (FSH) levels in the postmenopausal range. Until FSH is documented to be within menopausal range, treat the patient as WOCBP.
* Women ≥50 years old will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.

For randomisation at Visit 2b, patients should fulfil the following criteria:

1. ACQ-5 <1.5 at Visit 2b.
2. No increase (worsening) in ACQ-5 of at least ≥0.5 units between Visit 1 and Visit 2b compared to baseline.
3. No asthma exacerbation (see Section 8.1.3) between Visit 1 and Visit 2b.
4. No use of Ventolin® for symptom worsening in >3 out of the 7 days prior to Visit 2b.

Exclusion Criteria:

1. As judged by the Investigator, any evidence of a severe or serious treatment-related AE during Fasenra® treatment which in the Investigator's opinion makes it undesirable for the patient to participate in the study.
2. History of exacerbation requiring systemic corticosteroids or hospitalisation during the last 3 months prior to Visit 1 or during the run-in period.
3. Clinically important pulmonary disease other than asthma (eg, active lung infection, Chronic Obstructive Pulmonary Disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis), or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
4. Current smokers or former smokers with a smoking history ≥20 pack/years.
5. History of alcohol or drug abuse within 12 months prior to Visit 1.
6. A helminth parasitic infection diagnosed within 24 weeks prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.
7. History of anaphylaxis to any biologic therapy.
8. Known history of allergy or reaction to any component of the study treatment formulation.
9. A history of known immunodeficiency disorder, including history of a positive human immunodeficiency virus (HIV) test.
10. Current malignancy, or history of malignancy, except for:

    * Patients who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained.
    * Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.

    Prior/Concomitant Therapy
11. Oral corticosteroid use during the last 3 months prior to Visit 1.
12. Receipt of long-acting muscarinic antagonist (LAMAs) or theophyllines from Visit 1 until after Visit 8b, or leukotriene receptor antagonist (LTRAs) from Visit 2b until after Visit 8b.
13. Use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, or any experimental anti-inflammatory therapy) within 3 months or 5 half-lives (whichever is longer) prior to the date informed consent is obtained.
14. Receipt of live attenuated vaccines 30 days prior to Visit 1.
15. It is recommended to allow receipt of inactive/killed vaccinations (eg, inactive influenza) provided they are not administered within 1 week before/after any study treatment administration.
16. It is recommended to allow receipt of coronavirus disease 2019 (COVID-19) vaccination prior to study start provided such patients are not randomized until >30 days after last vaccine dose.
17. It is recommended to allow allergen immunotherapy provided it is stable for at least 30 days prior to Visit 1 and there is no anticipated change during the treatment period. Allergen immunotherapy should not be administered on the same day as study visits.
18. Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
19. Five-lipoxygenase inhibitors (eg, zileuton) are prohibited and are not allowed within 30 days of Visit 1 and until after Visit 8b.
20. Receipt of any marketed (eg, omalizumab) or investigational biologic within 4 months or 5 half-lives prior to the date informed consent is obtained, whichever is longer.
21. Receipt of systemic treatment with strong CYP3A4 inhibitors (eg, ketoconazole and itraconazole) from Visit 1 until after Visit 8b.
22. Receipt of beta-adrenergic blockers (including eye drops) from Visit 1 until after Visit 8b.
23. Concurrent participation in another clinical study with an Investigational Product or a post-authorisation safety study.

    Other Exclusions
24. Planned surgical procedures or other planned life events during the conduct of the study that would affect the patient's ability to comply with study treatment dosing or study assessments.
25. Involvement in the planning and/or conduct of the study (applies to both AZ staff and/or staff at the study site).
26. Judgement by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
27. Prior randomisation in the present study.
28. Currently pregnant, breast-feeding, or lactating women.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Jackson, Principal Investigator — Guy's & St Thomas' NHS Trust
Locations (22):
- France (6):
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Pessac
- Germany (9):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cottbus
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Jena
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, München
- Italy (3):
  - Research Site, Bergamo
  - Research Site, Napoli
  - Research Site, Roma
- United Kingdom (4):
  - Research Site, Belfast
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jackson DJ, Heaney LG, Humbert M, Kent BD, Shavit A, Hiljemark L, Olinger L, Cohen D, Menzies-Gow A, Korn S; SHAMAL Investigators. Reduction of daily maintenance inhaled corticosteroids in patients with severe eosinophilic asthma treated with benralizumab (SHAMAL): a randomised, multicentre, open-label, phase 4 study. Lancet. 2024 Jan 20;403(10423):271-281. doi: 10.1016/S0140-6736(23)02284-5. Epub 2023 Dec 7. PMID 38071986
- [Derived] Butler CA, Heaney LG. Fractional exhaled nitric oxide and asthma treatment adherence. Curr Opin Allergy Clin Immunol. 2021 Feb 1;21(1):59-64. doi: 10.1097/ACI.0000000000000704. PMID 33369570
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00072&attachmentIdentifier=5b51fe39-07bd-402c-9093-a83a7dc09f86&fileName=d3250c00072-study-synopsis+Errata_combined_with_Coverpage_Approved.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 27 July 2020 and 31 January 2023.
Pre-assignment Details: Study began with Screening Visit (Visit 1), followed by 4-8 weeks of screening and run-in. Patients previously exposed to benralizumab and ICS/LABA maintenance treatment prior to study entry received a high dose of Symbicort. At week 0 (Visit 2), 168 patients who met inclusion and randomization criteria were selected to participate in study and received study intervention benralizumab. These patients were randomly assigned to either treatment reduction arm or the reference arm.
Groups:
- Treatment Reduction: Patients received benralizumab 30 mg every 8 weeks (Q8W) during the study period, and high-dose Symbicort maintenance 400/12 μg ×2 inhalations BID + Ventolin (salbutamol 100 μg) reliever as needed (PRN), medium-dose Symbicort 200/6 μg ×2 inhalations BID maintenance + Symbicort 200/6 μg reliever PRN, low dose Symbicort 200/6 μg x 1 inhalation BID maintenance + Symbicort 200/6 μg reliever PRN; or Symbicort 200/6 μg reliever only, as per tapering scheme and depending on the degree of asthma control). The reduction period in this arm lasted for 32 weeks.
- Reference: Patients received benralizumab 30 mg Q8W + high-dose Symbicort® 400/12 μg maintenance × 2 inhalations BID + Ventolin® (salbutamol 100 μg) reliever PRN therapy. Eligible patients randomised to the reference arm continued on high-dose Symbicort® maintenance treatment and Ventolin® reliever treatment.
Period: Overall Study
Arm/Group | Treatment Reduction | Reference
Started | 125 | 43
Completed | 117 | 37
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Discontinued from study | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomised patients, irrespective of their protocol adherence and continued participation in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Reduction | Reference | Total
Number analyzed (Participants) | 125 | 43 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (12.44) | 56.5 (11.70) | 57.7 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 20 | 89
  Male | 56 | 23 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 91 | 28 | 119
  Unknown or Not Reported | 26 | 9 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95 | 31 | 126
  Asian | 0 | 2 | 2
  Other | 2 | 1 | 3
  Not Reported | 5 | 0 | 5
  Missing | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Reduced Their Symbicort® Maintenance Dose at the End of the Reduction Period
Description: Proportion of patients with non-missing Week 32 dose who reduced their Symbicort® maintenance dose at the end of the reduction period (Week 32) to: a) Medium-dose Symbicort® maintenance and reliever therapy (SMART), or b) Low-dose SMART, or c) Symbicort® anti-inflammatory reliever only.
Time Frame: At Week 32
Population: The FAS included all randomised patients, irrespective of their protocol adherence and continued participation in the study. Here, overall "number of participants analyzed" are the patients with available data that were evaluated for this outcome measure within the specified time frame.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Treatment Reduction
Number analyzed (Participants) | 119
Proportion of Participants
  Medium-dose SMART | 0.151 [0.0922 to 0.2285]
  Low-dose SMART | 0.168 [0.1058 to 0.2476]
  Symbicort® reliever-only dose | 0.605 [0.5113 to 0.6934]

2. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-5 Item (ACQ-5) Score at the End of the Reduction Period
Description: Change from baseline in the ACQ-5 patient reported outcome. This instrument contains 5 asthma symptom questions, rated from 0 (total control) to 6 (severely uncontrolled). The ACQ-5 score is the mean of the responses. Mean scores ≤0.75 indicate well controlled, scores between >0.75 and <1.5 indicate partly controlled, ≥1.5 indicate not well controlled asthma, and individual changes of ≥0.5 are considered to be clinically meaningful. ACQ-5 deterioration is defined as at least a 0.5 unit increase in ACQ-5 score from baseline, and a decrease of at least 0.5 units from baseline indicates improved asthma control.
Time Frame: Week 0 (baseline) and at Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 112 | 38
Score on a scale | 0.1617 (0.0393) | 0.0555 (0.0677)
Statistical Analysis 1: Comparison: Treatment Reduction vs Reference; Comparison with reference arm; Test type: Other — Mixed model for repeated measure (MMRM) with fixed effects for treatment arm, visit, baseline value, and treatment-by-visit interaction with an unstructured covariance structure; Least square mean difference = 0.1062, 95% CI 2-sided [-0.0485 to 0.2609]

3. Secondary Outcome: Change From Baseline in Standardised Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(S)+12) at the End of the Reduction Period
Description: The AQLQ(S)+12 is a Patient-Reported Outcome (PRO) that measures the health-related quality of life experienced by asthma patients. The questionnaire comprises 4 separate domains (symptoms, activity limitations, emotional function, and environmental stimuli). Patients are asked to recall their experiences during the previous 2 weeks before each visit and to score each of the questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). Range of Total Score = 0 - 7 as it is an average of responses to the individual questions. High score = better quality of life, and low score = poor quality of life. Change of >0.5 from baseline is considered a meaningful improvement in score.
Time Frame: Week 0 (baseline) and at Week 32
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 99 | 35
Score on a scale | -0.0279 (0.0559) | 0.0064 (0.0950)
Statistical Analysis 1: Comparison: Treatment Reduction vs Reference; Comparison with reference arm; Test type: Other — Comparison; Mixed model for repeated measure (MMRM); MMRM with fixed effects for treatment arm, visit, baseline value, and treatment-by-visit interaction with an unstructured covariance structure; Least square mean difference = -0.0343, 95% CI 2-sided [-0.2527 to 0.1841]

4. Secondary Outcome: Number of Patients With no Deterioration in AQLQ(S)+12 at the End of the Reduction Period
Description: The AQLQ(S)+12 is a PRO that measures the health-related quality of life experienced by asthma patients. The questionnaire comprises 4 separate domains (symptoms, activity limitations, emotional function, and environmental stimuli). Patients are asked to recall their experiences during the previous 2 weeks before each visit and to score each of the questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). AQLQ(S)+12 deterioration was defined as at least a 0.5 unit decrease in AQLQ(S)+12 total score from baseline. Patients with no deterioration include patients with improvement or no change.
Time Frame: At Week 32
Population: The FAS included all randomised patients, irrespective of their protocol adherence and continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 43
Participants
  Improvement | 12 | 3
  No change | 73 | 28

5. Secondary Outcome: Number of Patients With no Deterioration in ACQ-5 at the End of the Reduction Period
Description: Change from baseline in the ACQ-5 patient reported outcome. This instrument contains 5 asthma symptom questions, rated from 0 (total control) to 6 (severely uncontrolled). The ACQ-5 score is the mean of the responses. Mean scores ≤0.75 indicate well controlled, scores between >0.75 and <1.5 indicate partly controlled, ≥1.5 indicate not well controlled asthma, and individual changes of ≥0.5 are considered to be clinically meaningful. ACQ-5 deterioration is defined as at least a 0.5 units increase in ACQ-5 score from baseline, and a decrease of at least 0.5 units from baseline indicates improved asthma control.
Time Frame: At Week 32
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 43
Participants
  Improvement | 6 | 2
  No change | 87 | 28

6. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) During the Study Period
Description: The potential for benralizumab-treated patients to maintain lung function while stepping down Symbicort® maintenance treatment was assessed. The FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters. Change from baseline pre-bronchodilator FEV1 calculated as post-baseline pre-bronchodilator FEV1 (L) minus baseline pre-bronchodilator FEV1 (L) for all post-baseline measurement points.
Time Frame: At Week 0 (baseline), and at Weeks 8, 16, 24, 32, 40, and 48
Population: The FAS included all randomised patients, irrespective of their protocol adherence and continued participation in the study. Here, overall "number of participants analyzed", and "number analyzed" are the patients with available data that were evaluated for this outcome measure within the specified time frame.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 43
Liter
  Week 8: number analyzed (Participants) | 102 | 33
  Week 8 | 0.0411 (0.0183) | 0.0549 (0.0315)
  Week 16: number analyzed (Participants) | 97 | 34
  Week 16 | 0.0299 (0.0215) | 0.0115 (0.0363)
  Week 24: number analyzed (Participants) | 92 | 31
  Week 24 | -0.0536 (0.0317) | 0.0644 (0.0540)
  Week 32: number analyzed (Participants) | 89 | 31
  Week 32 | -0.0824 (0.0285) | -0.0016 (0.0482)
  Week 40: number analyzed (Participants) | 93 | 32
  Week 40 | -0.0953 (0.0280) | 0.0428 (0.0476)
  Week 48: number analyzed (Participants) | 92 | 29
  Week 48 | -0.0889 (0.0272) | 0.0059 (0.0475)

7. Secondary Outcome: Annualised Asthma Exacerbation Rate During the Study Period
Description: Asthma exacerbation rate was assessed. An asthma exacerbation was defined as a worsening of asthma symptoms that led to any of the following: a) Temporary bolus/burst of systemic corticosteroids (≥3 consecutive days); b) Single depo-injectable dose of corticosteroids (equivalent to a 3-day bolus/burst); c) Visit to emergency room/urgent care (treatment <24 hours) requiring systemic corticosteroids; d) Hospitalization (admission/evaluation ≥24 hours) due to asthma.
Time Frame: From Week 0 up to Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Events/Year
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 43
Events/Year | 0.14 [0.09 to 0.23] | 0.14 [0.06 to 0.31]

8. Secondary Outcome: Cumulative Total Daily Inhaled Corticosteroids (ICS) Dose, by Period
Description: The cumulative total daily ICS dose (maintenance +reliever) for: a) reduction period; b) maintenance period; c) study period was assessed.
Time Frame: Reduction period (From Week 0 up to Week 32); maintenance period (From Week 32 up to Week 48); Study period (Week 0 up to end of maintenance period/ end of study)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Microgram
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 42
Microgram
  Reduction period | 115956.8 (73223.93) | 312857.1 (81251.22)
  Maintenance period: number analyzed (Participants) | 102 | 38
  Maintenance period | 50984.3 (51148.59) | 150400.0 (42180.46)
  Study period | 157560.0 (114123.69) | 448933.3 (131247.22)

9. Secondary Outcome: Total Daily ICS Dose (Maintenance + Reliever) at the End of the Reduction Period
Description: The mean total daily ICS dose (maintenance + reliever) during the 8 weeks prior to end of the reduction period was assessed.
Time Frame: At Week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microgram
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 120 | 39
Microgram | 380.028 (440.4995) | 1401.796 (316.9718)

10. Secondary Outcome: Proportion of Participants Using the Same Symbicort® Daily Dose at the End of the Maintenance Period (Week 48) That They Achieved at the End of the Reduction Period (Week 32)
Description: Proportion of patients using the same Symbicort daily dose at the end of the maintenance period that they achieved at the end of the reduction period. Proportions were based on patients with non-missing Week 32 and Week 48 Symbicort doses.
Time Frame: At Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Treatment Reduction
Number analyzed (Participants) | 118
Proportion | 0.958 [0.9039 to 0.9861]

11. Secondary Outcome: Number of Patients With at Least 1 Exacerbation Occurring From End of the Reduction Period to End of the Maintenance Period
Description: Number of patients with at least 1 exacerbation occurring from end of the reduction period to end of the maintenance period.
Time Frame: From Week 32 to Week 48
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 43
Participants | 5 | 4

12. Secondary Outcome: Total Daily ICS Dose From the End of the Reduction Period to the End of the Maintenance Period
Description: Total daily ICS dose from the end of the reduction period to the end of the maintenance period.
Time Frame: Week 32, Week 40, and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Microgram
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 119 | 38
Microgram
  Week 32 | 383.221 (440.9649) | 1438.685 (220.6355)
  Week 40 | 408.458 (475.6986) | 1424.624 (321.5752)
  Week 48: number analyzed (Participants) | 117 | 38
  Week 48 | 376.356 (449.6614) | 1265.356 (472.5244)

13. Secondary Outcome: Change in ACQ-5 From the End of the Reduction Period to the End of the Maintenance Period
Description: Change in ACQ-5 score from end of reduction to end of maintenance is reported. This instrument contains 5 asthma symptom questions, rated from 0 (total control) to 6 (severely uncontrolled). The ACQ-5 score is the mean of the responses. Mean scores ≤0.75 indicate well controlled, scores between >0.75 and <1.5 indicate partly controlled, ≥1.5 indicate not well controlled asthma, and individual changes of ≥0.5 are considered to be clinically meaningful. ACQ-5 deterioration is defined as at least a 0.5 unit increase in ACQ-5 score from baseline, and a decrease of at least 0.5 units from baseline indicates improved asthma control.
Time Frame: From Week 32 to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 110 | 34
Score on a scale | -0.07 (0.575) | -0.20 (0.814)

14. Secondary Outcome: Change in AQLQ(S)+12 From the End of the Reduction Period to the End of the Maintenance Period
Description: Change in AQLQ(S)+12 from the end of the reduction period to the end of the maintenance period is reported. The AQLQ(S)+12 is a Patient-Reported Outcome (PRO) that measures the health-related quality of life experienced by asthma patients. The questionnaire comprises 4 separate domains (symptoms, activity limitations, emotional function, and environmental stimuli). Patients are asked to recall their experiences during the previous 2 weeks before each visit and to score each of the questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). Range of Total Score = 0 - 7 as it is an average of responses to the individual questions. High score = better quality of life, and low score = poor quality of life. Change of >0.5 from baseline is considered a meaningful improvement in score.
Time Frame: From Week 32 to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 97 | 31
Score on a scale | -0.008 (0.4720) | 0.060 (0.5658)

15. Secondary Outcome: Change in FEV1 From the End of the Reduction Period to the End of the Maintenance Period
Description: The change from the end of the reduction period to the end of the maintenance period for pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1) was calculated as Week 48 pre-bronchodilator FEV1 (Liter [L]) minus the maintenance period baseline pre-bronchodilator FEV1 (L). The FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration, expressed in liters.
Time Frame: From Week 32 to Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 100 | 30
Liter | 0.0089 (0.2320) | 0.0040 (0.2264)

16. Secondary Outcome: Number of Patients That Met Each Composite Endpoint Defining Clinical Remission
Description: The number of patients meeting each individual component of the composite endpoint defining clinical remission (zero exacerbations, ACQ-5 < 1.5, or ACQ-5 <= 0.75, < 10% FEV1 deterioration) at the end of reduction and maintenance periods were assessed.
Time Frame: At Week 32 and Week 48
Population: The FAS included all randomised patients, irrespective of their protocol adherence and continued participation in the study. Here, overall "number of participants analyzed" and "number analyzed" are the patients with available data that were evaluated for this outcome measure within the specified time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 119 | 38
Participants
  No asthma exacerbation at Week 32 | 108 | 37
  No asthma exacerbation at Week 48: number analyzed (Participants) | 117 | 37
  No asthma exacerbation at Week 48 | 101 | 32
  ACQ-5 <1.5 at Week 32: number analyzed (Participants) | 115 | 35
  ACQ-5 <1.5 at Week 32 | 106 | 32
  ACQ-5 <1.5 at Week 48: number analyzed (Participants) | 113 | 35
  ACQ-5 <1.5 at Week 48 | 103 | 32
  ACQ-5 ≤ 0.75 at Week 32: number analyzed (Participants) | 115 | 35
  ACQ-5 ≤ 0.75 at Week 32 | 65 | 21
  ACQ-5 ≤ 0.75 at Week 48: number analyzed (Participants) | 113 | 35
  ACQ-5 ≤ 0.75 at Week 48 | 68 | 21
  FEV1 < 10% decrease from baseline at Week 32: number analyzed (Participants) | 89 | 31
  FEV1 < 10% decrease from baseline at Week 32 | 59 | 26
  FEV1 < 10% decrease from baseline at Week 48: number analyzed (Participants) | 92 | 29
  FEV1 < 10% decrease from baseline at Week 48 | 66 | 23

17. Secondary Outcome: Number of Patients That Met 0, 1, 2, and All 3 Composite Remission Endpoints
Description: Clinical remission in patients at end of the reduction and maintenance periods was assessed. A remission score, assigning 1 point for each clinical remission component achieved at week 32 or week 48,was calculated for patients who met 0, 1, 2, and all 3 remission criteria (zero exacerbations,ACQ-5 < 1.5, or ACQ-5 <= 0.75,< 10% FEV1 deterioration). Total remission score ranges from 0 to 3. The higher the score, the more components of remission the patient achieved.
Time Frame: At Week 32 and Week 48
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 89 | 28
Participants
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 32: number analyzed (Participants) | 86 | 28
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 32: 0 | 2 | 0
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 32: 1 | 15 | 5
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 32: 2 | 40 | 8
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 32: 3 | 29 | 15
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 48: 0 | 1 | 1
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 48: 1 | 15 | 4
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 48: 2 | 41 | 9
  Remission score (Exacerbation, ACQ-5 ≤ 0.75, FEV1 < 10% decrease from baseline) at Week 48: 3 | 32 | 14
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 32: number analyzed (Participants) | 86 | 28
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 32: 0 | 1 | 0
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 32: 1 | 5 | 2
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 32: 2 | 32 | 5
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 32: 3 | 48 | 21
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 48: 0 | 0 | 0
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 48: 1 | 5 | 2
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 48: 2 | 36 | 7
  Remission score: Exacerbation, ACQ-5 < 1.5, FEV1 < 10% decrease from baseline at Week 48: 3 | 48 | 19

18. Secondary Outcome: Number of Patients With Adverse Events or Serious Adverse Events
Description: The safety and tolerability of benralizumab in patients with severe asthma, while stepping down Symbicort® maintenance treatment and maintaining asthma symptom control was assessed.
Time Frame: From Week 0 (randomization) to Week 48 or end of treatment (total period of study is 2.5 years)
Population: The safety analysis set (SAF) included all patients from the FAS who were randomized to the study and received any amount of study treatment during the ICS reduction and maintenance periods and used for all safety analyses. Here, overall "number of participants analyzed" are the patients with available data that were evaluated for this outcome measure within the specified time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Reduction | Reference
Number analyzed (Participants) | 125 | 42
Participants
  Any adverse event (AE) | 91 | 35
  Any AE with outcome = death | 0 | 0
  Any serious adverse event (including events with outcome = death) | 12 | 5
  Any AE leading to discontinuation of benralizumab | 3 | 1
  Any AE leading to discontinuation of Symbicort | 3 | 1
  Any AE leading to discontinuation of Ventolin | 2 | 1
  Any AE leading to withdrawal from study | 3 | 1

ADVERSE EVENTS:
Time Frame: Run-In period: Week -8 to -4 to Week 0 before randomization (total period of 8 weeks); Treatment Period (Treatment reduction and reference): From Week 0 (Randomization) to Week 48 or end of treatment (total period of study is 2.5 years)
Description: The safety analysis set (SAF) included all patients from the FAS who were randomized to the study and received any amount of study treatment during the ICS reduction and maintenance periods and used for all safety analyses. The run-in period includes adverse events occurring during this period reported by the patients in SAF.
Groups:
- Run-In Period: All patients at Screening (Visit 1), switched from their previous ICS/LABA maintenance treatment and rescue medication to high-dose Symbicort maintenance (budesonide/formoterol 400/12 μg) ×2 inhalations BID + Ventolin (salbutamol 100 μg) reliever PRN. Patients continued on this medication for the duration of the 4- to 8-week screening and run-in period.
Arm/Group | Run-In Period | Treatment Reduction | Reference
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/125 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/167 | 12/125 | 5/42
Other Adverse Events (participants affected / at risk) | 5/167 | 46/125 | 20/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Period (N=167) | Treatment Reduction (N=125) | Reference (N=42)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-In Period (N=167) | Treatment Reduction (N=125) | Reference (N=42)
Bronchitis (Infections and infestations) | 0 (0) | 7 (8) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 19 (19) | 9 (9)
Nasopharyngitis (Infections and infestations) | 3 (3) | 10 (12) | 7 (8)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 17 (20) | 4 (4)

LIMITATIONS AND CAVEATS:
In the CSR synopsis dated 11 September 2023, One patient was erroneously excluded from analysis. Correct count reveals 11 patients in the treatment reduction arm experienced at least one asthma exacerbation during treatment reduction period, resulting in a total of 11 exacerbations. As a consequence, analysis outputs for asthma exacerbation and remission have been affected, for which CSR errata have been submitted along with redaction package.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT04159519/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT04159519/SAP_001.pdf